CLINICAL TRIAL: NCT02581735
Title: Effectiveness of the uPatient Platform in the Fulfillment of the Prophylactic Treatment in Patients With Hemophilia
Brief Title: Effectiveness of the uPatient Platform in Prophylactic Treatment in Hemophilia
Acronym: uPatient
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Real Fundación Victoria Eugenia (Other)
Collaborators: Universidad de Murcia (Other); Medtep Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: uPatient
Record Dates: First submitted 2015-10-13; First posted 2015-10-21 (Estimated); Last update posted 2016-06-30 (Estimated); Status verified 2016-06

CONDITIONS: Haemophilia
Keywords: Haemophilia; Adherence; Prophylaxis treatment; Quality of Life; Illness Behavior; Veritas-Pro questionnaire; uPatient
MeSH Terms: conditions — Hemophilia A; Illness Behavior | interventions — hydroxyethyl methacrylate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with haemophilia: Using the platform Upatient, patients with hemophilia will register for one year, the prophylactic treatment who receive at home. Likewise, they indicate a replacement therapy as a result of joint bleeds.
  At baseline, a month, 6 months and at the end of the study, patients shall complete two questionnaires. The same way in the initial evaluation and end of the study, the clinical joint status will be evaluated with HJHS scale .
  Interventions: Other: Patients with haemophilia

INTERVENTIONS:
Other: Patients with haemophilia — Using the platform Upatient, patients with hemophilia will register for one year, the prophylactic treatment who receive at home. Likewise, they indicate a replacement therapy as a result of joint bleeds.
  At baseline, a month, 6 months and at the end of the study, patients shall complete two questionnaires. The same way in the initial evaluation and end of the study, the clinical joint status will be evaluated with HJHS scale .

SUMMARY:
Research project whose main objective is to evaluate the use of a technology platform (uPatient) to register the prophylactic treatment of patients with hemophilia treated in different Hematology and Hemotherapy services of several hospitals in Spain.

DETAILED DESCRIPTION:
The data obtained in this project will identify the level of compliance to the pharmacological treatment of patients with hemophilia prophylaxis. They will use different psychosocial questionnaires based on scientific evidence and the reliability of these, as well as its specific design for patients with hemophilia. Clinical data were also obtained regarding the joint of patients participating in the study state.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with hemophilia A or B
* Patients over 13 years old
* Patients on prophylactic treatment.

Exclusion Criteria:

* Patients who do not sign the informed consent document
* Patients who do not make domiciliary self-treatment
* Patients who do not have good adhesion to prophylactic treatment

Ages: 13 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with haemophilia
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Registration of the uPatient platform | Screening visit
  This register indicates the number of infusions
Change from baseline the quality of life at 6 months and at the end of the study | Screening visit, up to 4 weeks, up to 24 weeks and through study completion, an average of 1 year
  Quality of life questionnaire (SF-36)
Change from baseline the perception of disease at 6 months and at the end of the study | Screening visit, up to 4 weeks, up to 24 weeks and through study completion, an average of 1 year
  Questionnaire to evaluate the perception of disease (Questionnaire IPQ-R)
Change from baseline the compliance to the prophylactic treatment at 6 months and at the end of the study | Screening visit, up to 4 weeks, up to 24 weeks and through study completion, an average of 1 year
  Spanish version of the questionnaire for compliance to prophylactic treatment in patients with haemophilia (Veritas-Pro).
Change from baseline the joint status at the end of the study | Screening visit and through study completion, an average of 1 year
  Spanish version of the Haemophilia Joint Health Score (HJHS), to assess the joint status in patients with hemophilia

CONTACTS AND LOCATIONS:
Overall Officials: Rubén Cuesta-Barriuso, PhD, Principal Investigator — Real Fundación Victoria Eugenia